CLINICAL TRIAL: NCT05484921
Title: The Specificity and Sensitivity of circMETTL9 Gene in Patients With Traumatic Brain Injury, Its Correlation With Cognitive Function and Disturbance of Consciousness, and Prognosis
Brief Title: Clinical Significance of circMETTL9 Gene in Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-L129
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-04

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: traumatic brain injury; circMETTL9
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- traumatic brain injury group: (1) age 18-80 years, (2) admission due to isolated head injury, (3) unconsciousness at the time of injury. Isolated head trauma was defined as CT scan-confirmed brain injury without other major extracranial injuries, such as pelvis fractures, femur fractures, and severe invasive abdominal or thoracic injuries. Other exclusion criteria for patients were infection within the most recent month, previous head trauma, neurological diseases including ischemic and hemorrhagic stroke, use of antiplatelet or anticoagulant medications, and other prior systemic diseases including uremia, liver cirrhosis, malignancy, chronic heart disease, and chronic lung disease.

SUMMARY:
Objective: The relevance of circMETTL9 to the degree of injury, disturbance of consciousness, cognitive function and prognosis in patients with moderate to severe traumatic brain injury (TBI) remains unknown. The purpose of this study was to investigate the effect of circMETTL9 on the degree of injury, disturbance of consciousness, cognitive function and prognosis after TBI.

DETAILED DESCRIPTION:
1. Collect blood samples from patients with moderate to severe TBI and healthy people, and detect the expression of circMETTL9 by Real-time Quantitative PCR Detecting System(qPCR).Receiver operating characteristic curve (ROC) was used to analyze the sensitivity and specificity of circMETTL9 in TBI patients.
2. Using the Glasgow coma scale (GCS) and the coma recovery scale-revised (CRS-R) to assess the patient's disturbance of consciousness at 1, 3, 7, 14, and 21 days after TBI, respectively, The cognitive function of patients was assessed with the revised Rachel los amigos scale-revised (RLAS-R), and the correlation of circMETTL9 with disturbance of consciousness and cognitive function in TBI patients was analyzed.
3. Six months after TBI, the disability rating scale (DRS) and Glasgow outcome scale-extended (GOSE) were used to evaluate the prognosis of patients six months after discharge, and the correlation between circMETTL9 and prognosis was analyzed. sex.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years old, gender is not limited;
2. Have a clear history of TBI and be diagnosed by head CT, and it is the first episode;
3. Glasgow Coma Scale (GCS) score less than or equal to 12;
4. The condition is relatively stable, and there is no serious chronic disease;
5. Obtain informed consent from patients and (or) their families.

Exclusion Criteria:

1 Combined with severe underlying diseases such as respiratory failure, heart failure, liver and kidney insufficiency; previous stroke, intracranial tumor, intracranial infection, dementia, Alzheimer's disease, Parkinson's disease, endocrine disease, immune and blood system diseases.

2. Patients with pelvic fractures, substantial organ damage, etc., which may seriously affect the treatment effect at the time of injury;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TBI patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08-04 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of circMETTL9 in TBI patients were analyzed. | 2022-01-2023-12
  rComparison of serum cirMETTL9 expression levels among the three groups. The results of qRT-PCR showed that, compared with the healthy control group, the serum cirMETTL9 expression levels in the moderate TBI group and the severe TBI group were significantly increased, and the serum cirMETTL9 expression level in the severe TBI group was significantly higher than that in the patients with severe TBI. In the moderate TBI group, the difference was statistically significant (P < 0.05).

SECONDARY OUTCOMES:
The correlation of circMETTL9 in blood samples of TBI patients with disturbance of consciousness and cognitive function in TBI patients was analyzed. | 2022-01-2023-12
  Blood samples were collected from patients with moderate to severe TBI and healthy individuals, and the expression of circMETTL9 was detected by qPCR.
  Receiver operating characteristic curve (ROC) was used to analyze the sensitivity and specificity of circMETTL9 in TBI patients.

OTHER OUTCOMES:
The correlation between circMETTL9 and prognosis in blood samples of TBI patients was analyzed. | 2022-01-2023-12
  Six months after TBI, disability rating scale (DRS) and Glasgow outcome scale-extended (GOSE) were used to evaluate the prognosis of patients six months after discharge, and the correlation between circMETTL9 and prognosis was analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China